CLINICAL TRIAL: NCT03542461
Title: An Open-label, Randomized Phase III Study of Early Switch Maintenance vs DElayed Second-line Nivolumab in Advanced Stage Squamous Non Small-cell Lung Cancer (NSCLC) Patients After Standard First-line Platinum-based Chemotherapy - EDEN Trial
Brief Title: Early Switch Maintenance vs Delayed Second-line Nivolumab in Advanced Stage Squamous Non-small Cell Lung Cancer (NSCLC) Patients (EDEN Trial)
Acronym: EDEN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Mipharm S.p.A. (Unknown); Bioikos Ambiente Srl (Other); Istituto Toscano Tumori (Other); Temas srl (Unknown); Bristol Myers Squibb Srl Italia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-04-2016
Record Dates: First submitted 2018-03-05; First posted 2018-05-31 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Squamous Non-small Cell Lung Cancer
Keywords: Squamous NSCLC; Nivolumab
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Open-label, randomized in a 1:1 ratio to 2 treatment arms and stratified by centre and response to first-line induction therapy (minimization method)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A_Nivolumab (Experimental): Nivolumab 240 mg IV every 2 weeks until disease progression, unacceptable toxicity, patient refusal or Investigator's decision
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution
- B_Best Supportive Care (Other): Best Supportive Care until disease progression followed by Nivolumab at a dose of 240 mg IV until further disease progression, unacceptable toxicity, patient refusal or Investigator's decision.
  Interventions: Drug: Nivolumab 10 MG/ML Intravenous Solution; Other: Best Supportive Care

INTERVENTIONS:
Drug: Nivolumab 10 MG/ML Intravenous Solution — 240 mg as a 30 minutes IV infusion on Day 1 of each treatment cycle every 2 weeks, until intolerable toxicity or patient refusal or investigator's decision. In case of disease progression the treatment should be discontinued unless documented clinical benefits in the Investigator's judgement (no rapid progression, tolerance of trial drug, stable performance status, treatment maintenance does not delay an imminent intervention to prevent serious complication of PD) and no evidence of further progression at a radiographic assessment performed within 6 weeks. No dose escalations or reduction allowed. Administration delay until 6 weeks as well as resuming dose are allowed according to protocol defined criteria.
Other: Best Supportive Care — Care that aims to optimize the comfort, function and social support of the patients and their family at all stages of the illness. Best Supportive Care (BSC)includes the use of analgesics, antibiotics, blood tranfusions, blood products, radiotherapy, corticosteroids, antiemetics, antidiarrheals, vitamins and any intervention aiming the improvement of patient's discomfort. Any chemotherapy, immunotherapy and targeted therapy are not considered as part of BSC.
  Arms: B_Best Supportive Care

SUMMARY:
The study's hypothesis is that using Nivolumab as early switch maintenance, after 4-6 cycles of standard first-line chemotherapy, might improve survival in patients with advanced stage squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* pathologically (histology or cytology) confirmed diagnosis of squamous non-small cell lung cancer (NSCLC)
* histologically or cytologically confirmed stage IIIB-IV or recurrent squamous NSCLC with partial response (PR), complete response (CR) or stable disease (SD) according RECIST 1.1 after 4-6 courses of standard platinum-based chemotherapy (i.e. cisplatin or carboplatin combined with either paclitaxel, docetaxel, nab-paclitaxel, gemcitabine or vinorelbine)
* life expectancy ≥ 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PF) of 0-2
* last chemotherapy course completed within 8 weeks before randomization and radiological assessment for tumor evaluation after first-line chemotherapy within 4 weeks before randomization
* in case of presence of treated brain metastases, lesions should be stable for at least 4 weeks, steroids should be off or on stable dose (≤ 10 mg of prednisone or equivalent), radiotherapy should have been completed at least 14 days before randomization and any Adverse Event (AE) related to radiotherapy recovered to grade < 1 (except alopecia)
* in case of females: postmenopausal status (at least 12 months after last menstrual period should have been passed) before the screening visit or surgical sterilization. Women of childbearing potential (WOCBP) must use 2 effective methods of contraception (from the time of informed consent signature trough 30 days after last trial drug dose) or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. Pregnancy should be avoided for 23 weeks after the last trial drug dose. WOCBP must have negative serum or urine pregnancy test within 24 hours prior to the start of trial drug treatment.
* in case of males: even if surgically sterilized, effective barrier contraception (method with failure rate < 1%/year) during the entire study treatment period and for a period of 31 weeks after the last dose of trial drug, or practice true abstinence when this is in line with the preferred and usual lifestyle of the subject.
* laboratory parameters measured within 14 days prior randomization as follows: absolute neutrophil count ≥ 1000/mmc platelet count ≥ 75000/mmc haemoglobin ≥ 9g/dL total bilirubin ≤ 1.5x the Upper Normal Limit (local laboratory range) except in case of Gilbert Syndrome where total bilirubin value < 3.0 mg/dL is allowed serum alanine aminotransferase or aspartate aminotransferase or aspartate aminotransferase ≤ 3x the Upper Normal Limit (local laboratory range) creatinine ≤ 1.5x the Upper Normal Limit or estimated creatinine clearance using Cockcroft-Gault formula ≥ 30 mL/minute for patients with creatinine levels above institutional limits
* stable medical conditions, including the absence of acute exacerbations of chronic illnesses, serious infections or major surgery within 4 weeks before randomization and otherwise noted in other eligibility criteria
* ability to comply with protocol requirements
* ability to provide written informed consent

Exclusion Criteria:

* prior treatment with nivolumab or any other immunotherapy agent (e.g. anti-PD-1, anti-PD-L1, etc.)
* progressive disease after 4-6 cycles of first line platinum-based chemotherapy
* non-platinum-based first-line chemotherapy
* active, known or suspected autoimmune disease; please note: diabetes mellitus, hypothyroidism requiring only hormone replacement, skin disorders, such as vitiligo, psoriasis or alopecia, not requiring systemic treatment, or conditions not expected to recur without external trigger are not excluded.
* condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior randomization; please note: topical, ocular, intranasal and inhalational corticosteroids with minimal systemic absorption, adrenal replacement steroid doses > 10 mg/day prednisone equivalent without concurrent autoimmune disease, brief course of corticosteroids treatment or prophylaxis or treatment of non-autoimmune conditions are allowed.
* patients with symptomatic and/or progressive brain metastases or with carcinomatous meningitis.
* previous malignancies unless complete remission has achieved at least 2 years prior to the study entry and no additional therapy is required or anticipated during the study period
* any medical condition, within 6 months before receiving the first dose of trial drug, considered relevant in the investigator's opinion. Please note: chronic stable atrial fibrillation on stable anticoagulant therapy are not excluded. Pacemaker may represent an exclusion criterion and should be discussed with the project clinician. Attention should be paid to the conditions requiring treatment with potentially hepatotoxic drugs considering the hepatotoxic potential of the trial drug.
* infection requiring an antibiotic therapy or other serious infection within 14 days before the first dose of trial drug
* positive serum pregnancy test, pregnancy or breast feeding condition (only for females)
* major surgery within 4 weeks (or 2 weeks for minor surgery) before study enrollment and not fully recovered to baseline or to a stable clinical status; lease note: insertion of vascular device is not excluded.
* interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity known history of testing positive for Human Immunodeficiency Virus (HIV) or known acquired Immunodeficiency Syndrome (AIDS)
* any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* comorbidity or unresolved toxicities that would preclude administration of nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of death by any cause or study discontinuation due to lost to follow up/withdrawal of consent assessed up to 14 months .
  Time from randomization to death date. Please note: a subject who has not died will be censored at the last known date alive.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of the first documented tumor progression or death by any cause, whichever occurs first, assessed up to 6 months in the arm B and 10 months in arm A.
  Time from randomization to the date of the first documented tumor progression (RECIST 1.1) or death due to any cause. Please note: clinical deterioration not radiologically confirmed is not considered progression for the purpose of this measure. Subjects who did not have any study tumor assessments and did not die will be censored on the date they were randomized. Subjects who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last evaluable tumor assessment prior to the initiation od the subsequent anti-cancer therapy.
Progression-Free Survival from induction (PFSind) | From date of first chemotherapy cycle until the date of the first documented tumor progression or death for any cause, whichever occurs first, assessed up to 10 months in the arm B and 14 months in arm A.
  Time from first chemotherapy cycle until documented tumor progression or death by any cause.
Time to Treatment Failure (TTF) | From date of randomization until the date of treatment discontinuation, assessed up to 9 months in the arm B and 14 months in arm A.
  Time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patients preference, Investigator's decision or death.
Overall Survival from Induction (OSind) | From date of first chemotherapy cycle until the date of death, assessed assessed up to 14 months in the arm B and 18 months in arm A..
  Time from first chemotherapy cycle until death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ardizzoni, Dr, Principal Investigator — Medical Oncology Unit - S.Orsola Malpighi University Hospital of Bologna; Marcello Tiseo, Dr, Study Chair — Medical Oncology Unit - University Hospital of Parma
Locations (31):
- Italy (31):
  - UOC Oncologia - Azienda USL di Imola - Ospedale Santa Maria della Scaletta, Imola, Bologna
  - Oncologia Medica - IRST - IRCCS di Meldola, Meldola, Forlì
  - AUSL 12 Viareggio, Ospedale Versilia, Lido di Camaiore (LU) - Oncologia Medica, Lido di Camaiore, Lucca
  - UO Medicina Oncologica - Ospedale di Carpi (MO) - Azienda USL di Modena, Carpi, Modena
  - UOC di Oncologia Medica - ASST Valle Olona - Presidio Ospedaliero di Saronno, Saronno, Varese
  - SC Oncologia - ASO "SS Antonio e Biagio e Cesare Arrigo", Alessandria
  - UO Oncologia Medica - A.S.S.T. Papa Giovanni XXIII di Bergamo, Bergamo
  - UO di Oncologia Medica - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Divisione di Oncologia Medica - Ospedale di Bolzano, Bolzano
  - UOC Oncologia Medica - PO A.Perino ASL di Brindisi, Brindisi
  - SC di Oncologia - Istituti Ospitalieri di Cremona, Cremona
  - Dipartimento di Oncologia Medica - Azienda Ospedaliera S.Croce e Carle Cuneo - Ospedale Carle, Cuneo
  - UO di Oncologia Ematologia - Azienda Ospedaliero Universitaria di Ferrara, Ferrara
  - S.C. Oncologia Medica 1 - Azienda Ospedaliero Universitaria Careggi, Florence
  - UOS Tumori Polmonari - IRCCS AOU San Martino -IST- Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Azienda USL Toscana nord ovest - Ospedale San Luca di Lucca - Dipartimento Oncologico, Lucca
  - Azienda Ospedaliero-Universitaria di Modena - Policlinico - Dipartimento di Scienze Mediche e Chirurgiche, Materno Infantili e dell'adulto, Modena
  - SC di Oncologia Medica - A.O. San Gerardo, Monza
  - U.O.C Pneumologia ad Indirizzo Oncologico - AORN Ospedali dei Colli Monaldi, Napoli
  - IOV Istituto Oncologico Veneto - UOC di Oncologia Medica 2, Padua
  - UOC di Oncologia Medica - Azienda Ospedaliero Universitaria di Parma, Parma
  - S.C. di Oncologia Medica - Ospedale S.Maria della Misericordia, Perugia
  - AUSL - Piacenza - Ospedale "Guglielmo da Saliceto"-Dip.Oncologia e Ematologia- UO di Oncologia Medica Azienda, Piacenza
  - Azienda Ospedaliera Universitaria Pisana - Dipartimento Medico in Oncologia, Pisa
  - IRCCS CRO Aviano - SOC Oncologia medica e dei tumori Immunocorrelati - Dipartimento di Oncologia Pordenone S. Vito, Pordenone
  - Pneumologia ad Indirizzo Oncologico 1 - A.O. San Camillo Forlanini, Roma
  - Università la Sapienza - Policlinico Umberto I - Dipartimento di scienze radiologiche, oncologiche e anatomo-patologiche - UOC Oncologia B, Roma
  - UO Oncologia Medica - ASL N.1 di Sassari - Ospedale Civile di Sassari, Sassari
  - U.O. Oncologia Medica - Ospedale Santa Chiara, Trento
  - Reparto di Oncologia - Azienda Sanitaria Universitaria Integrata di Udine - Presidio Ospedaliero Santa Maria della Misericordia, Udine
  - U.S.O. GIVOP (Gruppo Interdisciplinare Veronese Oncologia Polmonare) Oncologia - Azienda Ospedaliera Integrata Verona, Verona

REFERENCES:
- [Background] Thatcher N, Hirsch FR, Luft AV, Szczesna A, Ciuleanu TE, Dediu M, Ramlau R, Galiulin RK, Balint B, Losonczy G, Kazarnowicz A, Park K, Schumann C, Reck M, Depenbrock H, Nanda S, Kruljac-Letunic A, Kurek R, Paz-Ares L, Socinski MA; SQUIRE Investigators. Necitumumab plus gemcitabine and cisplatin versus gemcitabine and cisplatin alone as first-line therapy in patients with stage IV squamous non-small-cell lung cancer (SQUIRE): an open-label, randomised, controlled phase 3 trial. Lancet Oncol. 2015 Jul;16(7):763-74. doi: 10.1016/S1470-2045(15)00021-2. Epub 2015 Jun 1. PMID 26045340
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Lilenbaum RC, Herndon JE 2nd, List MA, Desch C, Watson DM, Miller AA, Graziano SL, Perry MC, Saville W, Chahinian P, Weeks JC, Holland JC, Green MR. Single-agent versus combination chemotherapy in advanced non-small-cell lung cancer: the cancer and leukemia group B (study 9730). J Clin Oncol. 2005 Jan 1;23(1):190-6. doi: 10.1200/JCO.2005.07.172. PMID 15625373
- [Background] Stinchcombe TE, Choi J, Schell MJ, Mears A, Jones PE, Nachtsheim RV, Socinski MA. Carboplatin-based chemotherapy in patients with advanced non-small cell lung cancer and a poor performance status. Lung Cancer. 2006 Feb;51(2):237-43. doi: 10.1016/j.lungcan.2005.10.018. Epub 2005 Dec 27. PMID 16378657
- [Background] Zukin M, Barrios CH, Pereira JR, Ribeiro Rde A, Beato CA, do Nascimento YN, Murad A, Franke FA, Precivale M, Araujo LH, Baldotto CS, Vieira FM, Small IA, Ferreira CG, Lilenbaum RC. Randomized phase III trial of single-agent pemetrexed versus carboplatin and pemetrexed in patients with advanced non-small-cell lung cancer and Eastern Cooperative Oncology Group performance status of 2. J Clin Oncol. 2013 Aug 10;31(23):2849-53. doi: 10.1200/JCO.2012.48.1911. Epub 2013 Jun 17. PMID 23775961
- [Background] Paz-Ares LG, de Marinis F, Dediu M, Thomas M, Pujol JL, Bidoli P, Molinier O, Sahoo TP, Laack E, Reck M, Corral J, Melemed S, John W, Chouaki N, Zimmermann AH, Visseren-Grul C, Gridelli C. PARAMOUNT: Final overall survival results of the phase III study of maintenance pemetrexed versus placebo immediately after induction treatment with pemetrexed plus cisplatin for advanced nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Aug 10;31(23):2895-902. doi: 10.1200/JCO.2012.47.1102. Epub 2013 Jul 8. PMID 23835707
- [Background] Cappuzzo F, Ciuleanu T, Stelmakh L, Cicenas S, Szczesna A, Juhasz E, Esteban E, Molinier O, Brugger W, Melezinek I, Klingelschmitt G, Klughammer B, Giaccone G; SATURN investigators. Erlotinib as maintenance treatment in advanced non-small-cell lung cancer: a multicentre, randomised, placebo-controlled phase 3 study. Lancet Oncol. 2010 Jun;11(6):521-9. doi: 10.1016/S1470-2045(10)70112-1. Epub 2010 May 20. PMID 20493771
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Francisco LM, Sage PT, Sharpe AH. The PD-1 pathway in tolerance and autoimmunity. Immunol Rev. 2010 Jul;236:219-42. doi: 10.1111/j.1600-065X.2010.00923.x. PMID 20636820
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Background] Carter L, Fouser LA, Jussif J, Fitz L, Deng B, Wood CR, Collins M, Honjo T, Freeman GJ, Carreno BM. PD-1:PD-L inhibitory pathway affects both CD4(+) and CD8(+) T cells and is overcome by IL-2. Eur J Immunol. 2002 Mar;32(3):634-43. doi: 10.1002/1521-4141(200203)32:33.0.CO;2-9. PMID 11857337
- [Background] Barber DL, Wherry EJ, Masopust D, Zhu B, Allison JP, Sharpe AH, Freeman GJ, Ahmed R. Restoring function in exhausted CD8 T cells during chronic viral infection. Nature. 2006 Feb 9;439(7077):682-7. doi: 10.1038/nature04444. Epub 2005 Dec 28. PMID 16382236
- [Background] Dong H, Chen L. B7-H1 pathway and its role in the evasion of tumor immunity. J Mol Med (Berl). 2003 May;81(5):281-7. doi: 10.1007/s00109-003-0430-2. Epub 2003 Apr 30. PMID 12721664
- [Background] Konishi J, Yamazaki K, Azuma M, Kinoshita I, Dosaka-Akita H, Nishimura M. B7-H1 expression on non-small cell lung cancer cells and its relationship with tumor-infiltrating lymphocytes and their PD-1 expression. Clin Cancer Res. 2004 Aug 1;10(15):5094-100. doi: 10.1158/1078-0432.CCR-04-0428. PMID 15297412
- [Background] Thompson RH, Gillett MD, Cheville JC, Lohse CM, Dong H, Webster WS, Krejci KG, Lobo JR, Sengupta S, Chen L, Zincke H, Blute ML, Strome SE, Leibovich BC, Kwon ED. Costimulatory B7-H1 in renal cell carcinoma patients: Indicator of tumor aggressiveness and potential therapeutic target. Proc Natl Acad Sci U S A. 2004 Dec 7;101(49):17174-9. doi: 10.1073/pnas.0406351101. Epub 2004 Nov 29. PMID 15569934
- [Background] Mu CY, Huang JA, Chen Y, Chen C, Zhang XG. High expression of PD-L1 in lung cancer may contribute to poor prognosis and tumor cells immune escape through suppressing tumor infiltrating dendritic cells maturation. Med Oncol. 2011 Sep;28(3):682-8. doi: 10.1007/s12032-010-9515-2. Epub 2010 Apr 6. PMID 20373055
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651
- [Background] Brahmer JR, Drake CG, Wollner I, Powderly JD, Picus J, Sharfman WH, Stankevich E, Pons A, Salay TM, McMiller TL, Gilson MM, Wang C, Selby M, Taube JM, Anders R, Chen L, Korman AJ, Pardoll DM, Lowy I, Topalian SL. Phase I study of single-agent anti-programmed death-1 (MDX-1106) in refractory solid tumors: safety, clinical activity, pharmacodynamics, and immunologic correlates. J Clin Oncol. 2010 Jul 1;28(19):3167-75. doi: 10.1200/JCO.2009.26.7609. Epub 2010 Jun 1. PMID 20516446
- [Background] Gettinger SN, Horn L, Gandhi L, Spigel DR, Antonia SJ, Rizvi NA, Powderly JD, Heist RS, Carvajal RD, Jackman DM, Sequist LV, Smith DC, Leming P, Carbone DP, Pinder-Schenck MC, Topalian SL, Hodi FS, Sosman JA, Sznol M, McDermott DF, Pardoll DM, Sankar V, Ahlers CM, Salvati M, Wigginton JM, Hellmann MD, Kollia GD, Gupta AK, Brahmer JR. Overall Survival and Long-Term Safety of Nivolumab (Anti-Programmed Death 1 Antibody, BMS-936558, ONO-4538) in Patients With Previously Treated Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2015 Jun 20;33(18):2004-12. doi: 10.1200/JCO.2014.58.3708. Epub 2015 Apr 20. PMID 25897158
- [Background] Rizvi NA, Mazieres J, Planchard D, Stinchcombe TE, Dy GK, Antonia SJ, Horn L, Lena H, Minenza E, Mennecier B, Otterson GA, Campos LT, Gandara DR, Levy BP, Nair SG, Zalcman G, Wolf J, Souquet PJ, Baldini E, Cappuzzo F, Chouaid C, Dowlati A, Sanborn R, Lopez-Chavez A, Grohe C, Huber RM, Harbison CT, Baudelet C, Lestini BJ, Ramalingam SS. Activity and safety of nivolumab, an anti-PD-1 immune checkpoint inhibitor, for patients with advanced, refractory squamous non-small-cell lung cancer (CheckMate 063): a phase 2, single-arm trial. Lancet Oncol. 2015 Mar;16(3):257-65. doi: 10.1016/S1470-2045(15)70054-9. Epub 2015 Feb 20. PMID 25704439
- [Background] Pardoll D. Does the immune system see tumors as foreign or self? Annu Rev Immunol. 2003;21:807-39. doi: 10.1146/annurev.immunol.21.120601.141135. Epub 2001 Dec 19. PMID 12615893
- [Background] Zitvogel L, Tesniere A, Kroemer G. Cancer despite immunosurveillance: immunoselection and immunosubversion. Nat Rev Immunol. 2006 Oct;6(10):715-27. doi: 10.1038/nri1936. Epub 2006 Sep 15. PMID 16977338
- [Background] Dunn GP, Bruce AT, Ikeda H, Old LJ, Schreiber RD. Cancer immunoediting: from immunosurveillance to tumor escape. Nat Immunol. 2002 Nov;3(11):991-8. doi: 10.1038/ni1102-991. PMID 12407406
- [Background] Horne ZD, Jack R, Gray ZT, Siegfried JM, Wilson DO, Yousem SA, Nason KS, Landreneau RJ, Luketich JD, Schuchert MJ. Increased levels of tumor-infiltrating lymphocytes are associated with improved recurrence-free survival in stage 1A non-small-cell lung cancer. J Surg Res. 2011 Nov;171(1):1-5. doi: 10.1016/j.jss.2011.03.068. Epub 2011 Apr 22. PMID 21571304
- [Background] Al-Shibli KI, Donnem T, Al-Saad S, Persson M, Bremnes RM, Busund LT. Prognostic effect of epithelial and stromal lymphocyte infiltration in non-small cell lung cancer. Clin Cancer Res. 2008 Aug 15;14(16):5220-7. doi: 10.1158/1078-0432.CCR-08-0133. PMID 18698040
- [Background] Ruffini E, Asioli S, Filosso PL, Lyberis P, Bruna MC, Macri L, Daniele L, Oliaro A. Clinical significance of tumor-infiltrating lymphocytes in lung neoplasms. Ann Thorac Surg. 2009 Feb;87(2):365-71; discussion 371-2. doi: 10.1016/j.athoracsur.2008.10.067. PMID 19161739
- [Background] Greenwald RJ, Freeman GJ, Sharpe AH. The B7 family revisited. Annu Rev Immunol. 2005;23:515-48. doi: 10.1146/annurev.immunol.23.021704.115611. PMID 15771580
- [Background] Sharpe AH, Wherry EJ, Ahmed R, Freeman GJ. The function of programmed cell death 1 and its ligands in regulating autoimmunity and infection. Nat Immunol. 2007 Mar;8(3):239-45. doi: 10.1038/ni1443. PMID 17304234
- [Derived] Gelsomino F, Boni L, Tiseo M, Ricciardi S, Rocco D, Cortinovis DL, Proietto M, Cogoni A, Pasello G, Camerini A, Sperandi F, Colantonio I, Metro G, Mazzoni F, Baldini E, Veccia A, Bennicelli E, Cecilia Bettini A, Tognetto M, Ardizzoni A. An open-label, randomized phase III study of early switch maintenance vs delayed second-line nivolumab in advanced stage squamous non-small cell lung cancer (NSCLC) patients after standard first-line platinum-based chemotherapy-EDEN trial GOIRC 04-2016. Lung Cancer. 2025 Jan;199:108059. doi: 10.1016/j.lungcan.2024.108059. Epub 2024 Dec 15. PMID 39700681